CLINICAL TRIAL: NCT05248412
Title: The Long-term Spill-over Impact of COVID-19 on Health and Healthcare of Patients With Non-communicable Diseases (and Without COVID-19) : an In-depth Outcome and Health Economic Evaluation
Brief Title: The Long-term Spill-over Impact of COVID-19 on Health and Healthcare of People With Non-communicable Diseases
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, Chairperson of Department of Family Medicine & Primary Care, The University of Hong Kong
Other Study IDs: UW21-297
Record Dates: First submitted 2022-02-17; First posted 2022-02-21 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus; Hypertension; Cancer; Cardiovascular Diseases; Chronic Respiratory Disease; Kidney Disease, Chronic; Noncommunicable Diseases
Keywords: COVID-19 Pandemic; Morality; Complication; Utilization, Health Care; Noncommunicable Diseases
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Neoplasms; Cardiovascular Diseases; Renal Insufficiency, Chronic; Noncommunicable Diseases; COVID-19; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID-19 outbreaks — The intervention of the study is the COVID-19 outbreaks in Hong Kong. The pre-and post-COVID-19 outbreak periods will be defined as 1 January 2010 - 31 December 2019 and 1 January 2020 - 31 December 2024, respectively.

SUMMARY:
Objectives and aim: To evaluate the long-term spill-over (indirect) effect of Coronavirus disease (COVID-19) on health outcomes and healthcare utilization among people with non-communicable diseases and without COVID-19.

Design: A population-based cohort study using electronic health records of the Hospital Authority (HA) clinical management system, economic modeling, and serial cross-sectional surveys on healthcare service utilization.

Setting: HA public hospitals and outpatient clinics in Hong Kong

Participants: People aged ≥ 18 years with a documented diagnosis of diabetes mellitus, hypertension, cardiovascular disease, cancer, chronic respiratory disease, and chronic kidney disease; without COVID-19; attending HA services between 2010 and 2024.

Main outcome measures: All-cause mortality, disease-specific outcomes, healthcare service utilization, and costs.

Methods: The annual incidence of each outcome in each year between 2010 and 2024 will be calculated. An interrupted time-series analysis to assess the changes in outcomes between pre-and-post-COVID-19 outbreak periods. Long term health economic impact of healthcare disruptions during the COVID-19 outbreak will be modeled using microsimulation. Multivariable Cox proportional hazards regression and Poisson/negative binomial regression to evaluate the effect of different modes of care on the risk of the outcomes.

Implications: Findings will inform policies and practices on contingency care plans to avoid excessive morbidity and mortality and to assure the quality of care for patients with NCD as part of the territorial response to the health crisis.

DETAILED DESCRIPTION:
This study aims to evaluate the spill-over impact of the COVID-19 outbreak on health outcomes, healthcare utilization, and costs in patients with major non-communicable diseases (NCDs). The study will include six leading NCDs (diabetes mellitus, hypertension, cardiovascular diseases (CVD), cancer, chronic kidney diseases (CKD), chronic respiratory diseases) representing the most prevalent conditions and the major causes of deaths in Hong Kong. The objectives of the study are the following:

1. To determine changes in all-cause mortality, disease-specific outcomes, and healthcare utilization rates and costs among major NCD patients during the pre-and post- COVID-19 outbreak.
2. To assess the long-term health economic impact of COVID-19 on health outcomes and healthcare utilization rates and costs among major NCD patients by conducting an in-depth economic evaluation
3. To explore the impact of different modes of care on all-cause mortality, disease-specific outcomes, and healthcare utilization rates and costs among major NCD patients during the post-COVID-19 period.

This study consists of two study designs.

1. It is a retrospective cohort study using data extracted from the electronic medical records of the Hong Kong Hospital Authority (HA) Clinical Management System (CMS) from 1 January 2010 to 31 December 2024.

   * Anonymous data including socio-demographics, disease-specific parameters identified by International Classification of Primary Care, 2nd edition (ICPC-2) and the International Classification of Diseases, 9th revision, Clinical Modification (ICD-9-CM) will be extracted by the Hospital Authority statistics. There will be two phases of data extraction for the data collected in the periods 2010-2021 and 2022-2024.
2. The investigators will carry out two serial cross-sectional surveys on self-reported healthcare service utilization in the second and fourth years after the COVID-19 outbreak.

   * Two surveys will be conducted for patients with the major NCD recruited from outpatient clinics to collect data on healthcare service utilization patterns and rates in the years of 2020 and 2022 using a structured questionnaire.

ELIGIBILITY:
(For cohort study)

Inclusion Criteria:

* People aged 18 years or above with a documented doctor-diagnosed NCDs (diabetes mellitus, hypertension, cardiovascular disease, cancer, chronic kidney disease, or chronic respiratory disease )
* People who attended at least once HA hospitals, general or specialist out-patients clinics between 1 January 2010 and 31 December 2024

Exclusion Criteria:

- People with a documented doctor-diagnosed COVID-19

(For cross-sectional study)

Inclusion Criteria:

* People aged 18 years or above with a documented doctor-diagnosed NCDs (diabetes mellitus, hypertension, cardiovascular disease, cancer, chronic kidney disease, or chronic respiratory disease )
* All participants are able to communicate in either Chinese or English and provide informed consent.

Exclusion Criteria:

* People with a documented diagnosis of COVID-19 during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * People aged 18 years or above with documented doctor-diagnosed NCDs (diabetes mellitus, hypertension, cardiovascular disease, cancer, chronic kidney disease, or chronic respiratory disease).
  * People who attended at least once HA hospitals, general or specialist out-patients clinics during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Health outcomes | 5 years
  Incidence of all-cause mortality, and disease-specific complications (cardiovascular disease, end-stage renal disease, retinopathy, neuropathy and all-cause mortality) The disease are defined by the diagnosis codes International Classification of Primary Care, Second edition or International Classification of Diseases,Ninth Revision, Clinical Modification.

SECONDARY OUTCOMES:
Healthcare service utilization | 5 years
  Utilization rates and costs for public and private healthcare services including hospitalization (episodes, modes of admission and length of stay), specialist and general outpatient consultations (number of visits, modes of consultations, western/Chinese medicine), and Accident & Emergency Department (AED) attendances (triage urgency level for AED attendances at public hospital).

OTHER OUTCOMES:
Burden of diseases due to indirect effect of COVID-19 | 5 years
  Years of life lost (YLL), quality-adjusted life year (QALY), and disability-adjusted life year (DALY) attributable to delayed care resulting from the COVID-19 outbreak. Based on life expectancy for 10-year ages groups from the Census and Statistics Department life tables for 2017-19.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Family Medicine & Primary Care, LKS Faculty of Medicine, University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided